CLINICAL TRIAL: NCT03090516
Title: Clinical Study on Improving the Cognitive Function of Patients With Mild to Moderate Alzheimer's Disease by Using Ginkgo Biloba Dispersible Tablets
Brief Title: Clinical Efficacy of Ginkgo Biloba Extract in the Treatment of Alzheimer's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ting Wu, Director, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ginkgo biloba
Record Dates: First submitted 2017-03-04; First posted 2017-03-24 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Alzheimer's
Keywords: Ginkgo biloba dispersible tablets; Alzheimer's
MeSH Terms: interventions — Ginkgo Extract; Donepezil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A ：Donepezil (Experimental): A：People are randomly divided into three groups according to the educational conditiono，gender and age.
  Interventions: Drug: Donepezil
- Arm B ：Donepezil and Ginkgo biloba dispersible tablets (Experimental): B：People are randomly divided into three groups according to the educational conditiono，gender and age.
  Interventions: Drug: Ginkgo biloba dispersible tablets and Donepezil
- Arm C：Ginkgo biloba dispersible tablets (Experimental): C：People are randomly divided into three groups according to the educational conditiono，gender and age.
  Interventions: Drug: Ginkgo biloba dispersible tablets

INTERVENTIONS:
Drug: Ginkgo biloba dispersible tablets — Arm C：Ginkgo biloba dispersible tablets，0.15g at a time， three times a day.
  Other Names: Ginkgo biloba dispersible tablets and Donepezil;Donepezil
  Arms: Arm C：Ginkgo biloba dispersible tablets
Drug: Donepezil — Arm A：Aricept 5mg/day
  Other Names: Ginkgo biloba dispersible tablets;Ginkgo biloba dispersible tablets and Donepezil
  Arms: Arm A ：Donepezil
Drug: Ginkgo biloba dispersible tablets and Donepezil — Arm B：Ginkgo biloba dispersible tablets，0.15g at a time， three times a day.Aricept 5mg/day.
  Other Names: Donepezil;Ginkgo biloba dispersible tablets
  Arms: Arm B ：Donepezil and Ginkgo biloba dispersible tablets

SUMMARY:
This project explores Ginkgo biloba ester dispersible tablets influence on cognitive function in patients with mild-to-moderate elderly, to observe the effects of different intervention time on cognitive function, for alzheimer's patients in drug rehabilitation treatment provides an effective solution.

DETAILED DESCRIPTION:
The assessment of cognitive scales included Minimum Mental State Examination(MMSE), Alzheimer's Disease Assessment Scale-cognition(ADAS-cog), Neuropsychiatric inventory(NPI), quality of Life of Life in Alzheimer's disease(Qol-ADL), activities of Daily living(ADL), Geriatric Depression scale(GDS).Biochemical test included cholesterol, triglycerides, and low density lipoprotein.

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed with dementia caused by AD in 2011, the latest diagnostic criteria for Alzheimer's disease (NIA-AA), according to the patient's clinical and cranial imaging findings
2. Improved Hachinski ischemic scale score <4
3. All patients underwent head CT and / or MRI examinations and laboratory tests to rule out other causes of dementia
4. MMSE(High school≤24,Primary school≤20;illiteracy≤17)
5. CDR 1-2
6. The subjects and nurses signed informed consent, and the nursing staff were able to take responsibility for the supervision of the participants
7. The subjects were stable
8. Cooperate, willing to complete all parts of the research, and have the ability to complete the study alone or with the help of the nursing staff
9. To cooperate with the study, do not live alone, such as living alone should keep in touch with the nurse every day.

Exclusion Criteria:

1. Heart lung kidney disease, may interfere to evaluate the efficacy and safety of patients at risk or special disease,for example:Congestive heart failure et al.
2. According to NINDS-AIREN standard (Roman GC et al 1993) is currently diagnosed as possible vascular dementia
3. Improved Hachinski ischemic scale score（MHIS）≥4
4. Diagnosis of severe depression, schizophrenia, and other major neurodegenerative disorders, according to the DSM-IV axis
5. Neurological or other medical disorders that affect the function of the central nervous system,like Moderate anemia,Vitamin B12 or folic acid deficiency, et al. Not with the cognitive function examination (including blindness, deafness, severe language disorders).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-08-10 (Actual); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Scales to assess | change from baseline MMSE at 12weeks
  MMSE（Mini-mental State Examinatlon）
Electroencephalography P300 | change from baseline at 12weeks
  participants distinguish two voice and count them at the same time.we record their electroencephalography
liver function (blood) | change from baseline at 12weeks
  liver function（aspartate transaminase，Alanine aminotransferase，low density lipoprotein，Serum total cholesterol，Triglyceride）
1.5T MRI changes | changes before and after 12weeks
  Magnetic Resonance Imaging
Alzheimer disease assessment scale (ADAS-cog) | change from baseline ADAS-cog at 12 weeks
  ADAS-cog
activities of daily living scale (ADL) | change from baseline ADL at 12 weeks
  ADL
Change in neuropsychiatrc interventory (NPI) | change from baseline NPI at 12weeks
  NPI
Change in geriatric depression scale (GDS) | change from baseline GDS at 12 weeks
  GDS
renal function | change from baseline at 12weeks
  blood urea nitrogen

SECONDARY OUTCOMES:
ECG | change from baseline at 12weeks
  Electrocardiograph

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Ting Wu, Nanjing, Jiangsu, China